CLINICAL TRIAL: NCT00002814
Title: A Phase II Trial of Paclitaxel and Topotecan With Filgrastim in Patients With Recurrent or Refractory Glioblastoma Multiforme or Anaplastic Astrocytoma
Brief Title: Combination Chemotherapy for Patients With Brain Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9607; NCI-V96-0955 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — Filgrastim; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy using paclitaxel and topotecan, plus G-CSF, in treating patients with glioblastoma multiforme or anaplastic astrocytoma that is refractory or recurrent.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate in patients with refractory or recurrent glioblastoma multiforme or anaplastic astrocytoma treated with paclitaxel (TAX) and topotecan (TOPO) with granulocyte colony-stimulating factor (G-CSF) support. II. Determine survival in these patients. III. Describe the toxicity of TAX/TOPO/G-CSF. IV. Evaluate tumor p53 expression in relation to response to TAX/TOPO/G-CSF.

OUTLINE: All patients receive paclitaxel, topotecan, and G-CSF every 3 weeks for at least 2 courses and until 2 courses beyond maximum response. Patients are followed every 3 months for 2 years, then every 6 months for relapse and survival.

PROJECTED ACCRUAL: A total of 35 patients will be entered if there are 1-3 responses in the first 20 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Biopsy proven glioblastoma multiforme or anaplastic astrocytoma Central pathologic review at Dartmouth-Hitchcock Medical Center, including assay for tumor p53 expression No anaplastic oligodendroglioma No mixed oligodendroastrocytoma Recurrent or progressive disease following radiotherapy documented by CT or MRI within 2 weeks of entry

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60%-100% Hematopoietic: WBC at least 3,000 ANC at least 1,500 Platelets at least 100,000 Hepatic: Bilirubin no greater than 1.0 mg/dL AST/ALT no greater than 2.5 times normal Renal: Creatinine no greater than 1.5 mg/dL Other: No documented sensitivity to E. coli-derived products No major medical or psychiatric illness that would interfere with therapy or compliance with scheduled follow-up No pregnant or nursing women Adequate contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No prior taxanes or topoisomerase I inhibitors At least 4 weeks since chemotherapy (6 weeks since nitrosoureas) At least 4 weeks since radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 1996-08; Primary Completion 2001-04 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camilo E Fadul, MD, Study Chair — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States